CLINICAL TRIAL: NCT00587938
Title: BNP Measurement Reduces Resource Utilization for Patients With CHF Admitted Thorough the ED: A Clinical Development Project
Brief Title: BNP Measurement Reduces Resource Utilization for Patients With CHF Admitted Thorough the ED
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Dr Raquel Marie Schears MD, MPH, FACEP (Co-PI), Mayo Clinic
Other Study IDs: 1780-03
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-12

CONDITIONS: Congestive Heart Failure
Keywords: congestive heart failure; Brain naturietic peptide; hospital utilization cost
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Original protocol specifies a single 10 ml of blood is collected and frozen from each study participant (N=200), to be available for research assays.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: BNP level from protocol blood tests initiated in the ED, reported to ED physician prior to ED disposition.
- B: BNP level from protocol blood tests initiated in the ED, NOT reported to ED physician prior to ED disposition.

SUMMARY:
Measurement of brain natriuretic peptide (BNP) in dyspneic patients increases diagnostic accuracy for congestive heart failure (CHF). Limited information is available regarding economic outcomes attributable to BNP assay. The aim of this study was to assess the economic impact of BNP assay in elderly dyspneic patients presenting to the emergency department (ED).

DETAILED DESCRIPTION:
Dyspneic patients 65 years were enrolled in a randomized, controlled trial; hemodynamically unstable patients were excluded. BNP (Biosite assay) levels were measured prior to physician assessment with randomization in 1:1 ratio to either BNP 1) level reported or 2) level not reported. ED physicians made triage decisions guided by clinical judgment and nomogram to aid in interpretation of BNP level. Primary outcome was mean total hospital cost per subject. Secondary outcomes included admission rate, service assignment, discharge diagnosis and length of stay. Differences between groups were compared by t-test with bootstrap. Costs reflect 2005 constant dollars.

ELIGIBILITY:
Inclusion Criteria:

* Dyspneic patients 65 years or older presenting to the ED with chief complaint of shortness of breath.

Exclusion Criteria:

* hemodynamically unstability

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Dyspneic patients:65 years or older presenting to the ED with chief complaint of shortness of breath, were enrolled in a randomized, controlled trial.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2003-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Mean total hospital cost per subject | spans from ED eval through hospitalization discharge

SECONDARY OUTCOMES:
Included admission rate, service assignment, discharge diagnosis, and length of stay. | from ED evaluation through hospitalization discharge

CONTACTS AND LOCATIONS:
Overall Officials: Raquel M Schears, MD, MPH, Principal Investigator — Mayo Clinic; Alfredo L Clavell, MD, Principal Investigator — Mayo Clinic; Lyle J Olsen, MD, Study Chair — Mayo Clinic; Paula J Santrach, MD, Study Director — Mayo Clinic
Locations (1):
- Saint Marys Hospital, Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Schmidt TA, Salo D, Hughes JA, Abbott JT, Geiderman JM, Johnson CX, McClure KB, McKay MP, Razzak JA, Schears RM, Solomon RC; SAEM Ethics Committee. Confronting the ethical challenges to informed consent in emergency medicine research. Acad Emerg Med. 2004 Oct;11(10):1082-9. doi: 10.1197/j.aem.2004.05.028. PMID 15466152
- [Background] Clavell AL, Stingo AJ, Aarhus LL, Burnett JC Jr. Biological actions of brain natriuretic peptide in thoracic inferior vena caval constriction. Am J Physiol. 1993 Dec;265(6 Pt 2):R1416-22. doi: 10.1152/ajpregu.1993.265.6.R1416. PMID 8285286